# **Title**

Ketamine and/or lidocaine analgesia for abdominal surgery

# **Principal Investigator**

Rebecca Yuen Shi Wong, MBBS MPH

### **Co-Investigators**

Santiago Luis, MD Daniel Sessler, MD Jeffrey Jacobs, MD Edward Mascha, PhD Emanuele Lo Menzo, MD PhD Estelle Swanson, RN Rene Aleman, MD Joel Frieder, MD Ricardo Plata Aguilar, MD Gerges Azer, MD

### **INTRODUCTION**

Opioid overdoses cause 115 deaths per day in the United States, and cost more than \$500 billion in 2015, i.e. 2.8% of the nation's GDP (1). Concerningly, mortality due to the opioid epidemic has steadily increased with the number of deaths in 2016 being five times greater than in 1999 (2), and opioid prescribing having quadrupled in the same time frame (3).

The misuse of prescription opioids is reportedly the strongest risk factor for heroin abuse (3, 4), and in surgical patients, may have its roots in the perioperative period where over 80% are routinely exposed to opioids (5). Alam et al. reported a 44% increase in the risk of long-term opioid use in patients who were prescribed opioids after short-stay surgeries; even in opioid-naïve patients, an opioid prescription at hospital discharge was associated with 4.9 times the risk of chronic opioid use one year later (5). Thus, perioperative providers may be able to mitigate this threat by minimizing perioperative opioid use.

#### Background

Systemic lidocaine and ketamine are both analgesic agents, but by different mechanisms. The analgesic effects of intravenous lidocaine remain poorly characterized, but are thought to be related to its antiinflammatory effect and possibly blunted excitatory neuronal response (6). Ketamine is a NMDA antagonist, which has been implicated in nociception and the development of chronic pain (7).

Gilbert et al. first presented a case series in 1951 showing that an infusion of intravenous lidocaine markedly reduced pain in a wide spectrum of settings including cancer pain, postoperative pain, and labor pain (8). Following that, Ito and Ichiyanagi in 1974 showed that an infusion of a subanesthetic dose of ketamine also decreased postoperative pain after upper abdominal surgery (9). Many subsequent studies evaluated perioperative infusions of both agents; however, the doses and timings used across different types of surgery have been inconsistent, and the results have accordingly been variable (see Tables 1 and 2).

| Dose | Lidocaine (n = 23) | | Ketamine (n = 21) | |
|---|---|---|---|---|
| | Positive $(n = 17)$ | Negative $(n = 6)$ | Positive $(n = 16)$ | Negative $(n = 5)$ |
| Bolus | NO BOLUS (10) | NO BOLUS (27) | NO BOLUS (33) | 0.15 mg/kg (49) |
| | 100 mg (11-13) | 1.5 mg/kg (28-32) | 0.1 mg/kg (34) | 0.2 mg/kg(50) |
| | 1.5 mg/kg (14-23) | | 0.15 mg/kg (35-38) | 0.3 mg/kg (51) |
| | 2 mg/kg (24-26) | | 0.3 mg/kg (39-41) | 0.35 mg/kg (31) |
| | | | 0.5 mg/kg (42-47) | 0.4 m/kg (52) |
| | | | 1 mg/kg (48) | |
| Infusion | 2 mg/min for < 70 kg or 3 | 1 mg/min for $< 70$ kg or 2 | NO INFUSION (36-38, 44, | NO INFUSION (49, 51, 52) |
| | $mg/min for \ge 70 kg (19)$ | mg/min for $\geq 70 \text{ kg} (27)$ | 48) | 2.5 mcg/kg/min = 0.15 |
| | 2 mg/min (11, 12) | 2 mg/min (28) | 0.015 mg/kg/hr (33) | mg/kg/hr (50) |
| | 3 mg/min (13) | 2 mg/kg/hr (29, 31, 32) | 0.05 mg/kg/hr (41) | 0.2 mg/kg/hr (31) |
| | 1.5 mg/kg/hr (21, 22, 26) | 3 mg/kg/hr (30) | 2 mcg/kg/min = 0.12 mg/kg/hr | |
| | 2 mg/kg/hr (14-18, 20, 23, 25) | | (34, 35, 47) | |
| | 3 mg/kg/hr (10, 24) | | 3 mcg/kg/min = 0.18 mg/kg/hr | |
| | | | (39, 40) | |
| | | | 0.25 mg/kg/hr (42, 43) | |
| | | | 5 mcg/kg/min = 0.3 mg/kg/hr | |
| | | | (45) | |
| | | | 0.5 mg/kg/hr (46) | |

Table 1. Comparison of doses used in studies showing a positive versus negative effect on postoperative opioid consumption.

| Timing | Lidocaine (n = 23) | | Ketamine (n = 21) | |
|---|---|---|---|---|
| | Positive $(n = 17)$ | Negative $(n = 6)$ | Positive $(n = 16)$ | Negative $(n = 5)$ |
| Bolus | Before induction (13-17, 19, | Before induction (28-30) | Before induction (34, 37, 45) | Before induction (51) |
| | 25) | At induction (32) | At induction (39, 40, 43, 46) | After induction and before |
| | At induction (18, 20, 23) | After induction and before | After induction and before | incision (31, 49, 50, 52) |
| | After induction and before | incision (27, 31) | incision (33, 35, 36, 38, 41, 42, | |
| | incision (10-12, 21, 22, 24, 26) | | 44, 47, 48) | |
| Infusion | Until end of surgery (10, 16- | Until end of surgery (30) | Until end of surgery (34, 35, | 2.5 hr after incision (50) |
| | 18, 20, 23-26) | 4 hr postop (28) | 39-42, 45, 46) | 24 hr postop (31) |
| | 1 hr postop (19, 21, 22) | 24 hr postop (31, 32) | 48 hr postop (33, 43, 47) | |
| | 24 hr postop (11-15) | 48 hr postop (29) | | |
| | | 5 days postop or the day after | | |
| | | return of flatus (27) | | |

Table 2. Comparison of timings used in studies showing a positive versus negative effect on postoperative opioid consumption.

Disappointingly, Grady et al. did not show reduced 48-hour postoperative pain scores or opioid consumption with infusions of lidocaine with ketamine in patients recovering from open abdominal hysterectomy (31). Single preoperative doses of lidocaine and ketamine also did not reduce postoperative pain or opioid consumption after gynecological laparotomies (53). Conversely, ketamine has been found to reduce postoperative analgesic requirements as well as pain scores when used as an adjunct to lidocaine for intravenous regional anesthesia (54).

# Objective

We therefore propose to test the hypothesis that perioperative infusions of lidocaine and/or ketamine reduce opioid consumption and pain scores in adults recovering from elective inpatient abdominal surgery.

## **METHODS**

# Trial Design

We propose a prospective, randomized, double-blind, placebo-controlled clinical trial (RCT) with a factorial design

# **Participants**

We will include adults 18 to 80 years old having elective inpatient open or laparoscopic abdominal surgery with general anesthesia lasting 2 hours or longer.

#### Exclusion criteria:

- 1. Planned postoperative mechanical ventilation
- 2. Planned regional anesthesia/analgesia
- 3. Perioperative gabapentin, magnesium, or nitrous oxide use
- 4. Pregnancy or breastfeeding
- 5. Morbid obesity (BMI  $\geq$  35 kg/m<sup>2</sup>)
- 6. ASA physical status IV-V
- 7. Allergy to study medications
- 8. Contraindication to lidocaine (severe cardiac arrhythmia)
- 9. Contraindication to ketamine (psychiatric disorder, substance abuse, uncontrolled hypertension, pulmonary hypertension, increased intracranial or intraocular pressure, use of MAO inhibitors)
- 10. Chronic preoperative opioid use (> 90 morphine mg equivalents per day for > 3 months (55))
- 11. Significant preoperative hepatic dysfunction (ALT or AST > 5 times normal (56)) or planned liver transplantation
- 12. Preoperative cardiac failure (left ventricular ejection fraction  $\leq 40\%$  (57))
- 13. Unable to communicate or comprehend study instructions

# Interventions

- Patients will be given 1 g oral acetaminophen with a sip of water shortly before anesthetic induction.
- Patients will be factorially randomized to receive either lidocaine or placebo and either ketamine or placebo, resulting in the following four equal-sized groups:
  - Lidocaine + ketamine i.
  - ii. Lidocaine + placebo
  - iii. Ketamine + placebo

- iv. Placebo + placebo
- Blocked randomization (random sized) 1:1:1:1 will be based on computer-generated codes developed by Department of Outcomes Research statisticians. Allocation will be concealed until shortly before anesthetic induction with a web-based system that will record access and assignments.
- Lidocaine will be given as a 1.5 mg/kg bolus followed by an infusion of 2 mg/kg/hr based on actual body weight.
- Ketamine will be given as a 0.5 mg/kg/ bolus followed by an infusion of 0.3 mg/kg/hr based on actual body weight.
- Both the bolus and infusion will be started after induction and before incision.
- The infusion will be stopped one hour after transfer to PACU
- The boluses and infusions will be prepared by the pharmacy department, with normal saline as the placebo. Patients, anesthesiologists, and research fellows assessing the patients' postoperative outcomes will therefore all be blinded to the treatment group assignments.
- General anesthesia will be induced with propofol or etomidate and maintained with isoflurane. Intraoperative opioids will be restricted to only fentanyl.

### Measurements

Data to be collected includes:

- Baseline demographics: MRN, date of birth, gender (male/female), ethnicity, weight (kg) i.
- Surgery details: date of surgery, diagnosis, surgery, start case time (hr:min), end case time ii. (hr:min), intraoperative opioid (mg)
- Postoperative details: PACU discharge time (hr:min), hospital discharge time (date) iii.
- Total amount of perioperative lidocaine use (mg) iv.
- Total amount of perioperative ketamine use (mg) V.

The following will be measured at the end of the PACU stay as well as on the 1st and 2nd postoperative mornings:

- vi. Opioid consumption: preoperative (yes/no, type of opioid, average daily dose), postoperative (yes/no, type of opioid, cumulative dose from surgery to morning of POD2)
- vii. Pain scores: preoperative (0-10), postoperative (0-10)
- viii. Incidence of postoperative nausea or vomiting (yes/no)

Data that will be calculated from the aforementioned variables will include the following:

- Age (years) i.
- Surgery duration (hr:min) ii.
- iii. PACU length of stay (hr:min)
- Hospital length of stay (days) iv.
- Total amount of opioid consumption in PACU, POD1, and POD2 (oral morphine equivalent in V. mg)

Patient who are discharged before the 2<sup>nd</sup> POD will be contacted by phone for outcomes, and outpatient opioid consumption will be assessed by pill counts.

Data will be securely stored on the following: CCF's REDCap, CCF's shared network drives, CCF-issued computers, and CCF-issued encrypted USB drives. It may also be sent confidentially through the CCF email network. Results will be reported in an aggregate form and in a de-identified manner. The Cleveland Clinic Department of Outcomes Research will conduct the data analysis.

#### Outcomes

Joint primary outcome of:

- 1. Pain scores on a scale of 0-10/10, and
- 2. Total opioid consumption in oral morphine equivalents (mg) from the time of transfer to PACU through to the morning of POD2.
- The intervention will be deemed effective if both outcomes are non-inferior, and at least one is superior, to the control group.

### Secondary outcomes:

- 1. Overall benefit of analgesia score (OBAS)
- 2. Quality of recovery (OoR-15) score

All outcomes will be measured at the end of the PACU stay as well as on the 1st and 2nd postoperative mornings. On the 1<sup>st</sup> postoperative morning, patients will be asked to consider the period starting after discharge from the PACU. On the 2<sup>nd</sup> postoperative morning, patients will be asked to consider the period starting after the first postoperative morning.

Tertiary or exploratory outcomes

- 1. Time to first opioid administration (minutes)
- 2. Postoperative hospital length of stay (days)
- 3. Nausea or vomiting (yes/no)

The following adverse events will be monitored at the end of the PACU stay, on the morning of POD1 and the morning of POD2:

- Patient questionnaire: drowsiness, hallucination, peripheral neuropathy i (numbness/paresthesiae), tinnitus, nausea/vomiting
- ii. Nurse questionnaire: hypersensitivity reactions (rash, dyspnea, anaphylaxis), cardiac arrhythmia, confusion, seizure
- iii. Chart review: bradycardia/tachycardia (HR < 60 bpm or > 100 bpm), hypotension (SBP < 90 mmHg)

The trial will be managed by an Executive Committee consisting of Daniel I. Sessler, M. Alparslan Turan, and Edward J. Mascha.

### **Statistical Methods**

Randomized groups for each of the 2 factors (Lidocaine and Ketamine) will be compared on baseline variables using standardized difference. All analysis will be intent-to-treat.

# **Primary Outcomes**

Following the study aims, we define effectiveness of the analgesic agent (lidocaine or ketamine) for pain management as being noninferior to placebo on both pain control and opioid use, and at the same time being superior on either or both of pain control and opioid use. Therefore, we will first assess whether the agent (lidocaine or ketamine) is noninferior to placebo on each of pain score and opioid consumption. If the analgesic agent is found to be noninferior on both pain control and opioid use, we will then test whether the analgesic agent is superior over placebo on either pain control or opioid consumption, or both. We will first assess the treatment effects on each outcome, and then use those treatment effect estimates to test for noninferiority and superiority.

Pain score. The effects of lidocaine and ketamine, as well as their interaction, on the first primary outcome of pain score in the first 2 postoperative days will be assessed using a linear mixed effects model to adjust for the within-subject correlation on the pain scores over time. If there is a statistically significant (e.g., P<0.15) and clinically important (particularly, if effects are in opposite directions) interaction between the intervention factors on pain score, the interaction and confidence interval will be reported, and the main effects of each factor will be assessed within levels of the other factor. Otherwise, the main effects will be assessed collapsing over the other factor.

Opioid consumption. The effects of lidocaine and ketamine, as well as their interaction, on the second primary outcome of total opioid consumption through POD2 will be assessed using linear regression on the log-transformed values of the outcome, if appropriate. Otherwise, cumulative logit model or other appropriate method will be used to assess the main effects and their interaction. In the presence of a significant interaction, the main effects of each factor will be assessed within levels of the other factor. Otherwise, the main effects will be assessed collapsing over the other factor.

**Noninferiority**. For each analgesic agent (lidocaine and ketamine), we will test for noninferiority on pain score through a one-sided test using the treatment effect estimates and standard errors from the above linear mixed effects model and using a noninferiority delta of 1 point. We will test for noninferiority on opioid consumption using 1-tailed t-test on log-transformed opioid consumption (if appropriate – see above methods), using a noninferiority delta of 0.18 (log-scale equivalent of a ratio of 1.2 in geometric means). Noninferiority will be assessed at the overall 0.025 significance level for each agent, and using the same 0.025 as the significance criterion for each outcome within each agent. No adjustment for multiple testing will be needed since noninferiority is required on both outcomes for an agent (intersection-union test).

**Superiority.** Superiority test on pain control and opioid use will be performed only when the analgesic agent is noninferior to placebo on both pain score and opioid consumption. One-sided tests using the estimated treatment effects and standard errors and a significance criterion of 0.025/2=0.0125 will be used, adjusting for the fact that significance on either outcome would be sufficient to claim "superiority".

# **Secondary Outcome**

We will assess the effect of lidocaine and ketamine, as well as their interaction on OBAS and total QoR-9/QoR-15 scores through linear regression model.

### **Tertiary Outcome**

For time to first opioid administration and hospital length of stay, the two variables will be transformed to meet model assumptions of normality. We will then assess the effect of lidocaine and ketamine, as well as their interaction through linear regression model.

For nausea or vomiting at the end of PACU stay, POD1 and POD2, we will then assess the effect of lidocaine and ketamine, as well as their interaction through a generalized mixed effect model to account for within-subject correlation (random effect for subject) and the binary outcome type.

#### **Interim Analyses.**

Interim analyses will be done at each 25% of the planned maximum enrollment to assess for efficacy and futility using a group sequential design with gamma spending functions, and using gamma of -4 for efficacy and -1 for futility for each intervention. With this design, and assuming the hypothesized

treatment effects (25% reduction in opioid consumption, 2 points in pain score), the cumulative probability of crossing an efficacy or futility boundary at the 1st, 2nd, 3rd or 4th look will be 0.09, 0.40, 0.78, 1.00, respectively.

SAS 9.4 statistical software, Carey, NC, and R statistical software version 3.5.1 for 64-bit Windows operating system (The R Foundation for Statistical Computing, Vienna, Austria) will be used for all analyses.

# Sample Size

We base the sample size calculations on being able to claim either lidocaine or ketamine to be effective, and assuming no interaction between the two interventions. Based on the records we have for patients who went through colorectal surgery, opioid consumption through POD2 is approximately lognormally distributed. From these records, we observed means (SD) for pain scores to be 5 (2) and 4 (2), respectively for POD1 and POD2. Total opioid consumption for POD1 and POD2 has a mean (SD) of 257 (186), for an estimated coefficient of variation of 0.72.

We assume similar variability in pain scores and coefficient of variation for opioid consumption for the current study. Sample size calculation is based on 90% power to detect a difference in pain score of 2 points (out of 10) and 25% reduction in mean of opioid consumption with an overall significance level of 0.025 for each outcome. Sample size is driven by opioid consumption. Total sample size needed to detect a 25% reduction in opioid consumption is 272, 420 and 568, respectively, for coefficient of variance of 0.75, 1, and 1.25, adjusting for 2 outcomes (i.e., using significance criterion of 0.0125).

We will assume a CV of 1.0 to begin the study, and re-evaluate the CV during the trial, at the first interim analysis. If a larger CV is estimated, the sample size will be appropriately increased, with no statistical penalty. Therefore, before interim monitoring adjustment a total of 420 patients are needed. With interim monitoring adjustment, a total of 476 is needed.

#### **HUMAN SUBJECTS**

Lidocaine and ketamine are both medications commonly used in patient care with well-established safety profiles, as can be seen in previous studies.

We propose to charge the cost of the study medications to study participants as this treatment regimen is currently used in our institution on a routine basis, with 20 out of 23 anesthesiologists (87%) affirming its use for postoperative analgesia. The project should therefore not require any funding sources.

Consent will be obtained at least a day before surgery in the preoperative surgical or anesthesia clinics, where the discussion will be conducted by the research fellows in conjunction with the surgeon or anesthesiologist interviewing the patient.

### **REFERENCES**

- The Council of Economic Advisers. The underestimated cost of the opioid crisis. Washington, D.C.: Executive Office 1. of the President of the United States; 2017 Nov [cited 2018 Jul 22]. Available from: https://www.whitehouse.gov/sites/whitehouse.gov/files/images/The%20Underestimated%20Cost%20of%20the%20Opioid%20 Crisis.pdf.
- 2. Centers for Disease Control and Prevention. Understanding the Epidemic | Drug Overdose | CDC Injury Center. Atlanta, GA: U.S. Department of Health & Human Services; 2017 Aug 30 [cited 2018 Jul 22]. Available from: https://www.cdc.gov/drugoverdose/epidemic/index.html.
- Rudd RA, Aleshire N, Zibbell JE, Gladden RM, Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morbidity and mortality weekly report. 2016;64(50-51):1378-82.
- Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths United States, 2010-2015. MMWR Morbidity and mortality weekly report. 2016:65(5051):1445-52.
- Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesthesia and analgesia. 2017;125(5):1733-40.
- Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, et al. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. The Cochrane database of systematic reviews. 2018;6:Cd009642.
- Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA surgery. 2017;152(7):691-7.
- Gilbert CR, Hanson IR, Brown AB, Hingson RA, Intravenous use of xylocaine. Current researches in anesthesia & analgesia, 1951:30(6):301-13.
- 9. Ito Y, Ichiyanagi K. Post-operative pain relief with ketamine infusion. Anaesthesia. 1974;29(2):222-6.
- 10. Wu CT, Borel CO, Lee MS, Yu JC, Liou HS, Yi HD, et al. The interaction effect of perioperative cotreatment with dextromethorphan and intravenous lidocaine on pain relief and recovery of bowel function after laparoscopic cholecystectomy. Anesthesia and analgesia. 2005;100(2):448-53.
- Cassuto J, Wallin G, Hogstrom S, Faxen A, Rimback G. Inhibition of postoperative pain by continuous low-dose intravenous infusion of lidocaine. Anesthesia and analgesia. 1985;64(10):971-4.
- Wallin G, Cassuto J, Hogstrom S, Linden I, Faxen A, Rimback G, et al. Effects of lidocaine infusion on the sympathetic response to abdominal surgery. Anesthesia and analgesia. 1987;66(10):1008-13.
- Rimback G, Cassuto J, Tollesson PO. Treatment of postoperative paralytic ileus by intravenous lidocaine infusion. Anesthesia and analgesia. 1990;70(4):414-9.
- Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, et al. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007;106(1):11-8; discussion 5-6.
- Tikuisis R, Miliauskas P, Samalavicius NE, Zurauskas A, Samalavicius R, Zabulis V. Intravenous lidocaine for postoperative pain relief after hand-assisted laparoscopic colon surgery; a randomized, placebo-controlled clinical trial. Techniques in coloproctology. 2014;18(4):373-80.
- Lauwick S, Kim DJ, Michelagnoli G, Mistraletti G, Feldman L, Fried G, et al. Intraoperative infusion of lidocaine reduces postoperative fentanyl requirements in patients undergoing laparoscopic cholecystectomy. Canadian journal of anaesthesia = Journal canadien d'anesthesie. 2008;55(11):754-60.
- Yang SY, Kang H, Choi GJ, Shin HY, Baek CW, Jung YH, et al. Efficacy of intraperitoneal and intravenous lidocaine on pain relief after laparoscopic cholecystectomy. The Journal of international medical research. 2014;42(2):307-19.
- Song X, Sun Y, Zhang X, Li T, Yang B. Effect of perioperative intravenous lidocaine infusion on postoperative recovery following laparoscopic Cholecystectomy-A randomized controlled trial. International journal of surgery (London. England). 2017;45:8-13.
- Groudine SB, Fisher HA, Kaufman RP, Jr., Patel MK, Wilkins LJ, Mehta SA, et al. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesthesia and analgesia. 1998;86(2):235-9.
- Lauwick S, Kim DJ, Mistraletti G, Carli F. Functional walking capacity as an outcome measure of laparoscopic prostatectomy; the effect of lidocaine infusion. British journal of anaesthesia. 2009;103(2):213-9.
- Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, et al. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesthesia and analgesia. 2004;98(4):1050-5, table of contents.
- Baral BK, Bhattarai BK, Rahman TR, Singh SN, Regmi R. Perioperative intravenous lidocaine infusion on postoperative pain relief in patients undergoing upper abdominal surgery. Nepal Medical College journal: NMCJ. 2010;12(4):215-20.
- De Oliveira GS, Jr., Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesthesia and analgesia, 2012;115(2):262-7.
- Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, et al. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. British journal of anaesthesia. 2006;97(5):640-6.

- 25. Saadawy IM, Kaki AM, Abd El Latif AA, Abd-Elmaksoud AM, Tolba OM. Lidocaine vs. magnesium: effect on analgesia after a laparoscopic cholecystectomy. Acta anaesthesiologica Scandinavica. 2010;54(5):549-56.
- 26. Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesthesia and analgesia. 2009;109(5):1464-9.
- 27. Swenson BR, Gottschalk A, Wells LT, Rowlingson JC, Thompson PW, Barclay M, et al. Intravenous lidocaine is as effective as epidural bupivacaine in reducing ileus duration, hospital stay, and pain after open colon resection: a randomized clinical trial. Regional anesthesia and pain medicine. 2010;35(4):370-6.
- 28. Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, et al. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Annals of surgery. 2007;246(2):192-200.
- 29. Wongyingsinn M, Baldini G, Charlebois P, Liberman S, Stein B, Carli F. Intravenous lidocaine versus thoracic epidural analgesia: a randomized controlled trial in patients undergoing laparoscopic colorectal surgery using an enhanced recovery program. Regional anesthesia and pain medicine. 2011;36(3):241-8.
- 30. Bryson GL, Charapov I, Krolczyk G, Taljaard M, Reid D. Intravenous lidocaine does not reduce length of hospital stay following abdominal hysterectomy. Canadian journal of anaesthesia = Journal canadien d'anesthesie. 2010;57(8):759-66.
- 31. Grady MV, Mascha E, Sessler DI, Kurz A. The effect of perioperative intravenous lidocaine and ketamine on recovery after abdominal hysterectomy. Anesthesia and analgesia. 2012;115(5):1078-84.
- 32. Wuethrich PY, Romero J, Burkhard FC, Curatolo M. No benefit from perioperative intravenous lidocaine in laparoscopic renal surgery: a randomised, placebo-controlled study. European journal of anaesthesiology. 2012;29(11):537-43.
- 33. Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active-and placebo-controlled clinical trial. Minerva anestesiologica. 2016;82(10):1069-76.
- 34. Snijdelaar DG, Cornelisse HB, Schmid RL, Katz J. A randomised, controlled study of peri-operative low dose s(+)-ketamine in combination with postoperative patient-controlled s(+)-ketamine and morphine after radical prostatectomy. Anaesthesia. 2004;59(3):222-8.
- 35. Guignard B, Coste C, Costes H, Sessler DI, Lebrault C, Morris W, et al. Supplementing desflurane-remifentanil anesthesia with small-dose ketamine reduces perioperative opioid analgesic requirements. Anesthesia and analgesia. 2002;95(1):103-8, table of contents.
- 36. Roytblat L, Korotkoruchko A, Katz J, Glazer M, Greemberg L, Fisher A. Postoperative pain: the effect of low-dose ketamine in addition to general anesthesia. Anesthesia and analgesia. 1993;77(6):1161-5.
- 37. Kwok RF, Lim J, Chan MT, Gin T, Chiu WK. Preoperative ketamine improves postoperative analgesia after gynecologic laparoscopic surgery. Anesthesia and analgesia. 2004;98(4):1044-9, table of contents.
- 38. Kafali H, Aldemir B, Kaygusuz K, Gursoy S, Kunt N. Small-dose ketamine decreases postoperative morphine requirements. European journal of anaesthesiology. 2004;21(11):916-7.
- 39. Lee MH, Chung MH, Han CS, Lee JH, Choi YR, Choi EM, et al. Comparison of effects of intraoperative esmolol and ketamine infusion on acute postoperative pain after remifentanil-based anesthesia in patients undergoing laparoscopic cholecystectomy. Korean journal of anesthesiology. 2014;66(3):222-9.
- 40. Choi SK, Yoon MH, Choi JI, Kim WM, Heo BH, Park KS, et al. Comparison of effects of intraoperative nefopam and ketamine infusion on managing postoperative pain after laparoscopic cholecystectomy administered remifentanil. Korean journal of anesthesiology. 2016;69(5):480-6.
- 41. Sen H, Sizlan A, Yanarates O, Emirkadi H, Ozkan S, Dagli G, et al. A comparison of gabapentin and ketamine in acute and chronic pain after hysterectomy. Anesthesia and analgesia. 2009;109(5):1645-50.
- 42. De Kock M, Lavand'homme P, Waterloos H. 'Balanced analgesia' in the perioperative period: is there a place for ketamine? Pain. 2001;92(3):373-80.
- 43. Bicer F, Eti Z, Saracoglu KT, Altun K, Gogus FY. Does the Method and Timing of Intravenous Ketamine Administration Affect Postoperative Morphine Requirement After Major Abdominal Surgery? Turkish journal of anaesthesiology and reanimation. 2014;42(6):320-5.
- 44. Singh H, Kundra S, Singh RM, Grewal A, Kaul TK, Sood D. Preemptive analgesia with Ketamine for Laparoscopic cholecystectomy. Journal of anaesthesiology, clinical pharmacology. 2013;29(4):478-84.
- 45. Yalcin N, Uzun ST, Reisli R, Borazan H, Otelcioglu S. A comparison of ketamine and paracetamol for preventing remifentanil induced hyperalgesia in patients undergoing total abdominal hysterectomy. International journal of medical sciences. 2012;9(5):327-33.
- 46. Kararmaz A, Kaya S, Karaman H, Turhanoglu S, Ozyilmaz MA. Intraoperative intravenous ketamine in combination with epidural analgesia: postoperative analgesia after renal surgery. Anesthesia and analgesia. 2003;97(4):1092-6, table of contents
- 47. Zakine J, Samarcq D, Lorne E, Moubarak M, Montravers P, Beloucif S, et al. Postoperative ketamine administration decreases morphine consumption in major abdominal surgery: a prospective, randomized, double-blind, controlled study. Anesthesia and analgesia. 2008;106(6):1856-61.
- 48. Papaziogas B, Argiriadou H, Papagiannopoulou P, Pavlidis T, Georgiou M, Sfyra E, et al. Preincisional intravenous low-dose ketamine and local infiltration with ropivacaine reduces postoperative pain after laparoscopic cholecystectomy. Surgical endoscopy. 2001;15(9):1030-3.

- 49. Aubrun F, Gaillat C, Rosenthal D, Dupuis M, Mottet P, Marchetti F, et al. Effect of a low-dose ketamine regimen on pain, mood, cognitive function and memory after major gynaecological surgery: a randomized, double-blind, placebo-controlled trial. European journal of anaesthesiology. 2008;25(2):97-105.
- 50. Katz J, Schmid R, Snijdelaar DG, Coderre TJ, McCartney CJ, Wowk A. Pre-emptive analgesia using intravenous fentanyl plus low-dose ketamine for radical prostatectomy under general anesthesia does not produce short-term or long-term reductions in pain or analgesic use. Pain. 2004;110(3):707-18.
- 51. Kotsovolis G, Karakoulas K, Grosomanidis V, Tziris N. Comparison between the combination of gabapentin, ketamine, lornoxicam, and local ropivacaine and each of these drugs alone for pain after laparoscopic cholecystectomy: a randomized trial. Pain practice: the official journal of World Institute of Pain. 2015;15(4):355-63.
- 52. Dahl V, Ernoe PE, Steen T, Raeder JC, White PF. Does ketamine have preemptive effects in women undergoing abdominal hysterectomy procedures? Anesthesia and analgesia. 2000;90(6):1419-22.
- 53. Garcia-Navia JT, Tornero Lopez J, Egea-Guerrero JJ, Vilches Arenas A, Vazquez Gutierrez T. Effect of a single dose of lidocaine and ketamine on intraoperative opioids requirements in patients undergoing elective gynecological laparotomies under general anesthesia. A randomized, placebo controlled pilot study. Farmacia hospitalaria: organo oficial de expresion cientifica de la Sociedad Espanola de Farmacia Hospitalaria. 2016;40(1):44-51.
- 54. Abdel-Ghaffar HS, Kalefa MA, Imbaby AS. Efficacy of ketamine as an adjunct to lidocaine in intravenous regional anesthesia. Regional anesthesia and pain medicine. 2014;39(5):418-22.
- Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain United States, 2016. MMWR Recommendations and reports: Morbidity and mortality weekly report Recommendations and reports. 2016;65(1):1-49.
- 56. Kwo PY, Cohen SM, Lim JK. ACG Clinical Guideline: Evaluation of Abnormal Liver Chemistries. The American journal of gastroenterology. 2017;112(1):18-35.
- 57. Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE, Jr., Drazner MH, et al. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Journal of the American College of Cardiology. 2013;62(16):e147-239.